CLINICAL TRIAL: NCT06892782
Title: Effect of Hot Pack Application on Gastrointestinal Motility After Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Talhaoglu, assistant professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: hot pack in abdominal surgery
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hot Water Pack Application (Experimental): Patients in the intervention group will receive hot water pack application to the lumbar region. After the surgery, a hot water pack (heated to 40-42°C) will be applied to the lumbar region of the patient for 20 minutes, three times a day during the first 48 postoperative hours. The goal is to assess the effect of this intervention on gastrointestinal motility, including the time to first postoperative gas, first stool, and initiation of oral intake.
  Interventions: Other: Hot Water Pack Application
- Routine Care (No Intervention): Patients in the control group will receive routine postoperative care as per standard clinical practices. This group will not receive hot water pack application, and will instead undergo the usual procedures followed in the postoperative period to support recovery after abdominal surgery.

INTERVENTIONS:
Other: Hot Water Pack Application — A hot water pack heated to 40-42°C will be applied to the lumbar region of the patient for 20 minutes at three intervals per day during the first 48 hours post-surgery.
  Arms: Hot Water Pack Application

SUMMARY:
Study Title:

The Effect of Hot Water Pack Application to the Lumbar Region on Gastrointestinal Motility in Postoperative Abdominal Surgery Patients

Study Type:

Interventional (Randomized Controlled Trial)

Study Design:

Allocation: Randomized Intervention Model: Parallel Assignment Masking: Single-blind (Outcome Assessor) Primary Purpose: Supportive Care

Condition:

Postoperative Gastrointestinal Motility in Abdominal Surgery Patients

Interventions:

Experimental: Hot Water Pack Application Intervention: Application of a hot water pack (heated to 40-42°C) to the lumbar region for 20 minutes, three times a day, in the first 48 postoperative hours.

Purpose: To evaluate its effect on gastrointestinal motility and postoperative recovery.

Control: Routine Care Intervention: Standard postoperative care without hot water pack application.

Primary Outcome Measures:

Time to First Postoperative Gas (Hours) [Time Frame: Up to 72 hours]

Time to First Postoperative Stool (Hours) [Time Frame: Up to 72 hours] Time to Initiation of Oral Intake (Hours) [Time Frame: Up to 72 hours]

Secondary Outcome Measures:

Incidence of Postoperative Nausea and Vomiting (PONV) [Time Frame: Up to 72 hours] Severity of Abdominal Distension [Time Frame: Up to 72 hours]

Quality of Recovery-15 (QoR-15) Scale Score [Time Frame: Postoperative Days 1 and 3]

Gastrointestinal Symptom Rating Scale (GSRS) Score [Time Frame: Postoperative Days 1 and 3]

Eligibility Criteria:

Inclusion Criteria:

Abdominal surgery in the general surgery ward Age ≥ 18 years BMI between 18.50-24.99 kg/m² Able to communicate verbally Conscious, oriented, and willing to participate

Exclusion Criteria:

Previous gastrointestinal surgery Postoperative complications History of small bowel resection, ileostomy, or colostomy History of inflammatory bowel disease, emergency surgery, neoadjuvant therapy, appendectomy Chronic opioid use Chronic constipation (≤ 2 bowel movements per week) Abdominal radiotherapy ICU admission or postoperative bleeding

Estimated Enrollment:

80 participants (40 intervention, 40 control)

DETAILED DESCRIPTION:
This study is a randomized controlled experimental design aimed at evaluating the effect of hot water pack application to the lumbar region on gastrointestinal motility (time to first postoperative gas, first stool, and initiation of oral intake) in patients undergoing abdominal surgery. The study will be conducted in the postoperative period.

Participants

The study will include patients who undergo abdominal surgery in the general surgery ward. Participants will be randomly assigned to one of two groups:

Intervention Group (Hot Water Pack Application) Control Group (Routine Care) Interventions

Intervention Group (Hot Water Pack Application):

Procedure: A hot water pack will be applied to the lumbar region for 20 minutes, three times a day during the first 48 postoperative hours. The hot water packs will be heated to a temperature of 40-42°C.

Purpose: To assess its effect on postoperative gastrointestinal motility (e.g., first gas, first stool, initiation of oral intake).

Control Group (Routine Care):

Procedure: Participants will receive standard postoperative care, which includes usual practices for abdominal surgery recovery without hot water pack application.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older

Undergoing elective surgery

ASA I and III (American Society of Anesthesiologists physical status classification)

In the postoperative period, pulse, blood pressure, and body temperature within normal limits

Patients without previous gastrointestinal system surgery

Exclusion Criteria:

Previous gastrointestinal tract surgery

Complications in the postoperative period

History of small bowel resection and ileostomy or colostomy

History of inflammatory bowel diseases, emergency surgery, neoadjuvant therapy, appendectomy surgery

Chronic opioid use

Experiencing chronic constipation (≤ 2 bowel movements per week)

Receiving abdominal radiotherapy

Patients admitted to intensive care unit and patients with bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
bowel motility | postoperative 1-3 day
  Gastrointestinal Symptom Rating Scale (GSRS) - Scale Scores The Gastrointestinal Symptom Rating Scale (GSRS) is a validated tool used to assess the severity of gastrointestinal (GI) symptoms. It consists of 15 items, each scored on a 7-point Likert scale (1 = no discomfort, 7 = severe discomfort).
  Scoring Interpretation:
  Total Score Range: 15 to 105 (higher scores indicate worse GI symptoms). Mean score calculation: Total score is divided by the number of items (15) to determine the severity of symptoms.
  GSRS Subdimensions:
  The GSRS evaluates five symptom clusters:
  Reflux (2 items) → Heartburn, regurgitation Abdominal pain (3 items) → Stomach pain, hunger pain, nausea Indigestion (4 items) → Bloating, burping, early satiety, stomach rumbling Diarrhea (3 items) → Loose stools, urgency, frequency Constipation (3 items) → Hard stools, straining, incomplete evacuation
  Interpretation of Scores:
  15 - 30 → Mild symptoms 31 - 60 → Moderate symptoms 61 - 105 → Severe symptoms